CLINICAL TRIAL: NCT00111423
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety of Extended Treatment With Pegsunercept (PEG sTNF-RI) in Subjects With Rheumatoid Arthritis (RA)
Brief Title: Evaluating the Safety of Extended Treatment With Pegsunercept (PEG sTNF-RI)in Subjects With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20020133
Record Dates: First submitted 2005-05-20; First posted 2005-05-23 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, Inflammation; Pegsunercept, PEG sTNF-RI; Autoimmune, Amgen; Clinical Trials
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation | interventions — PEGylated soluble tumor necrosis factor receptor I

INTERVENTIONS:
Drug: Pegsunercept (PEG sTNF-RI)

SUMMARY:
The purpose of this study is to evaluate the safety of an additional 28 weeks of treatment with pegsunercept for subjects who have completed treatment in a previous double-blind study (20000201 or 20000198). In addition, this study will evaluate the efficacy and the feasibility of subject self-administration on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria: - Subjects who have completed 24 weeks of double-blind treatment in a previous protocol (20000201 or 20000198) - Females of childbearing potential and males must practice adequate contraception, in the judgement of the investigator, during the course of the study - The subject or legally acceptable representative must give informed consent for participation in the study before any study specific procedures are performed Exclusion Criteria: - Greater than a 7-day duration from the week 24 visit in the previous study to the first dose in this study - Any medical disability or condition (e.g., evidence of clinically significant liver dysfunction, active infection requiring treatment with systemic anti-infective agents) that would interfere with the assessment of safety of the study material or would compromise the ability of the subject to provide adequate informed consent - Concurrent treatment with an investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216
Dates: Start 2002-08

PRIMARY OUTCOMES:
Treatment-emergent adverse events

SECONDARY OUTCOMES:
Description of RA assessment outcomes
Assessment of Compliance

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20020133.pdf